CLINICAL TRIAL: NCT01486212
Title: Ischemia-reperfusion Injury Model on Healthy Volunteers and Measurement of Oxidative and Inflammatory Markers
Acronym: IROX-NH
Status: Completed | Type: Observational
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Natalie Løvland Halladin, M.D., Herlev Hospital
Other Study IDs: IROX-NH
Record Dates: First submitted 2011-11-17; First posted 2011-12-06 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-12

CONDITIONS: Ischemia-reperfusion Injury
Keywords: Ischemia-reperfusion injury; Oxidative markers; Inflammatory markers
MeSH Terms: conditions — Reperfusion Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy volunteers.: Male aged 18-40 years. Non-smokers. No known familiar disposition to vascular/heart diseases. No intake of prescription medicine.

SUMMARY:
Oxygen is necessary for the survival of oxygen consuming organisms. But the organisms metabolism alter the oxygen to free radicals. Free radicals are molecules which due to their structure can react with other molecules resulting in cell damage. This damage is due to several mechanisms.

This is e.g what happens when human tissue is cut of from blood supply for a time, and the blood supply is again restored. The damage following the restoration of blood is known as "ischemia-reperfusion injury". The reopening of the vessels and thereby supplying oxygenated blood to the deprived tissue can in it self contribute to cell death due to excessive amounts of free radicals. Antioxidants can neutralize free radicals and thereby minimize their damage.

The purpose of the investigators methodology study is to make an ischemia-reperfusion model on healthy volunteers (on the lower limb) to examine the expression of markers that are expressed in the muscle and the blood when blood supply is cut of to an area and later restored. The investigators wish to measure the product of the damage caused by free radicals and the levels of antioxidants.

If the investigators can produce elevation of oxidative and inflammatory markers, this model can be used to test antioxidative intervention.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Between 18 and 40 years.
* Non smokers.
* No known history of familiar cardio/vascular diseases.
* No intake of prescription medicine.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers. Male aged 18-40 years. Non smokers. No known history of familiar cardio/vascular diseases. No intake of prescription medicine.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2011-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Malondialdehyde (MDA) in muscle. | A change from baseline to 30 minutes after ischemia.
  Malondialdehyde (MDA), is a direct product of the lipidperoxidation occuring during reperfusion. It is caused by damage done by the free radicals.

SECONDARY OUTCOMES:
Malondialdehyde (MDA) in blood | A change from baseline measured in blood to 5, 15, 30, 60 and 90 minutes after reperfusion.
Vitamin C | A change from baseline measured in blood to 5, 15, 30, 60 and 90 minutes after reperfusion.
  Vitamin C is an antioxidant.
YKL-40 | A change from baseline measured in blood to 5, 15, 30, 60 and 90 minutes after reperfusion.
  YKL-40 is a marker that become elevated if local inflammation occurs.
Cytokines (Interleukin 1β,4,6,10 og TNF-α) | A change from baseline measured in blood to 5, 15, 30, 60 and 90 minutes after reperfusion.
  Interleukin (IL)- 1β, IL-6 og TNF-α are pro-inflammatory markers. IL-4 og IL-10 are anti-inflammatory markers.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Halladin, MD, Principal Investigator — Herlev Hospital
Locations (1):
- Herlev Hospital, Herlev, Herlev, Denmark